CLINICAL TRIAL: NCT06822426
Title: A Phase 3, Prospective, Multicenter, Double-Blind, Randomized, Controlled, Adaptive Study To Demonstrate The Safety And Efficacy Of DEFENCATH® In Reducing Central Line-Associated Bloodstream Infections (CLABSIs) In Adult Participants Receiving Total Parenteral Nutrition (TPN) Via Central Venous Catheter (CVC)
Brief Title: Comparing The Safety And Efficacy Of DEFENCATH® In Reducing Central-Line Bloodstream Infections (CLABSIs) In Adults Receiving Total Parenteral Nutrition Through A Central Venous Catheter (CVC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CorMedix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NUTRI-GUARD
Expanded Access: NCT06707480 (Available)
Record Dates: First submitted 2025-01-15; First posted 2025-02-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Central Line Associated Blood Stream Infections (CLABSI)
MeSH Terms: interventions — taurolidine; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DefenCath® (Experimental)
  Interventions: Drug: (taurolidine and heparin) catheter lock solution
- Control (Active Comparator)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: (taurolidine and heparin) catheter lock solution — for central venous catheter installation use
  Arms: DefenCath®
Drug: Heparin — Heparin
  Arms: Control

SUMMARY:
This is a Phase 3, randomized, double-blind, controlled, adaptive, 2-arm, multicenter study to demonstrate the efficacy and safety of DefenCath in adult participants receiving home Total Parenteral Nutrition (TPN) via Central Venous Catheter (CVC) compared with heparin.

ELIGIBILITY:
1. Participants who are resident within the US and Türkiye.
2. Participants who are male or female, aged ≥18 years at the time of consent.
3. Participants must sign and provide informed consent.
4. Participants who have a permanent tunneled CVC or permanent peripherally inserted central catheter (PICC) made of silicone or polyurethane, which has been in place for at least 7 days prior to enrollment.
5. Participants who require long-term (>6 months) TPN based on the investigator assessments.
6. Participants who require TPN for at least 3 days per week, of which 2 days have to be parenteral nutrition (PN).
7. Participants who have a minimum of a 4-hour CLS dwelling time and are willing to lock all lumens at a minimum of every 7 days.
8. Participants who are clinically stable, in the opinion of the investigator, for at least 4 weeks prior to enrollment.
9. Participants who are able and willing to be trained or have a caregiver who is willing and able to be trained on the instillation, aspiration of DefenCath or heparin, and to maintain a daily diary.
10. Male or female participants:

    1. Women of childbearing potential (WOCBP; see Section 4.5.1) must have a negative pregnancy test at screening (i.e., the participant is not pregnant); not be lactating; and use an acceptable method of contraception including but not limited to, abstinence, bilateral tubal ligation, vasectomized partner, a barrier method (diaphragm or condom), Depo-Provera, intrauterine device, or hormonal contraceptive (oral, implant, ring, patch) for the duration of the program until at least 30 days after the last DefenCath CLS instillation. (NOTE: The participant must have used the chosen method of birth control for at least 1 month/cycle prior to enrollment into the study).
    2. Male participants who are sexually active with a female partner of childbearing potential must agree to use male condoms with spermicide, even if the male participant has undergone a successful vasectomy (males with vasectomy can use condoms without spermicide), from Day 1 until at least 30 days after the last DefenCath CLS instillation.
11. Participants who comply with all study procedures and follow-up evaluations.

Exclusion Criteria:

1. Any participant unable or not willing to sign inform consent.
2. Any participant who has received systemic antibiotic within the last 14 days. Topical antibiotics are permitted. Use of metronidazole or rifaximin for treating small intestinal bacterial overgrowth (SIBO) is also permitted.
3. Any participant with visible evidence of compromised skin integrity present at the catheter exist site or catheter exit site infection.
4. Any participant with temporary, non-tunneled CVC or temporary PICC.
5. Any participant that has received thrombolytic treatment (e.g., tissue-type plasminogen activator [tPA]-Cathflo), not as a part of the institution's standard of care for patency management, in current catheter within 30 days of randomization.
6. Any participant with unstable arrhythmia, defined as presence of hemodynamic instability within a month prior to the baseline assessment.
7. Any participant using any type of antimicrobial-coated or heparin-coated catheter.
8. Any participant with documented chronic bleeding diathesis, active or recurrent bleeding within 1 month prior to randomization.
9. Any participant with a congenitally lethal condition or a life expectancy of less than 6 months.
10. Any participant with documented history of an atrial thrombus or known hypercoagulable state.
11. Any participant with an open, non-healing skin ulcer.
12. Any participant who has received a bone marrow transplant (allogeneic or autogenic/autologous) within the last year.
13. Any participant with neutropenia with an absolute neutrophil count <1000 cells/μL
14. Any participant with current requirement for systemic immunosuppression that would increase risk of infection including, but not limited to:

    1. Steroid use at an equivalent dose of prednisone 20 mg/day anticipated or actual for at least 8 weeks.
    2. Systemic chemotherapy.
    3. Methotrexate dose sufficiently high to suppress white blood cell count (WBC) count below 5,000 cells/μL.
    4. Azathioprine dose greater than 2.5 mg/kg/day.
    5. Calcineurin inhibitors:

    i. Cyclosporine dose greater than 8 mg/kg. ii. Tacrolimus dose greater than 0.4 mg/kg. f. Sirolimus dose greater 10 mg/daily.
15. Any participant with known allergies or absolute contraindications to citrate, taurolidine, or heparin or a history of heparin-induced thrombocytopenia.
16. Any participant taking other medication with known systemic drug interaction with citrate, taurolidine or heparin.
17. Any participant anticipating receiving a transplant within 90 days. Participants can be on a transplant list but a participant with a known or anticipated transplant date within 90 days of study entry should be excluded from study participation. A participant who may receive a transplant >90 days of study entry may remain on the study as long as they continue to receive TPN.
18. Any participant who is pregnant or lactating.
19. Any participant receiving continuous TPN (infusion over 24 hours).
20. Any participant with any medical conditions that render them unable to, or unlikely to complete the study or would interfere with optimal participation in the study or produce significant risk to participant.
21. Any participants who are participating in another interventional clinical study, except for non-pharmacological research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between treatment groups of proportion of participants who experience a Central Line-Associated Bloodstream Infections (CLABSI) within 12 months of the start of the study | Self-administered by participants (or a designated caregiver) per the participants regular TPN/ line access schedule, through study completion (up to 12 months)
  The proportion of participants who remain infection-free in the treatment groups will be compared, censoring participants who do not experience a CLABSI within 9 months, but fail to complete the 12 month follow-up period of the study.

SECONDARY OUTCOMES:
Incidence of AEs, SAEs, treatment-emergent adverse events (TEAEs) | Self-administered by participants (or a designated caregiver) per the participants regular TPN/ line access schedule, through study completion (up to 12 months)
  Compare the safety profile of DefenCath for use as a Catheter Lock Solution (CLS) in adult participants receiving Total Parenteral Nutrition (TPN) through a Central Venous Catheter (CVC) to the control of heparin CLS
Incidence of changes in laboratory evaluations, vital signs, or physical exam findings | Self-administered by participants (or a designated caregiver) per the participants regular TPN/ line access schedule, through study completion (up to 12 months)
  Compare the safety profile of DefenCath for use as a CLS in adult participants receiving TPN through a CVC to the control of heparin CLS

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of California Los Angeles, Los Angeles, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Bioresearch Partner, Doral, Florida
  - Emory University Hospital - GCRC, Atlanta, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Johns Hopkins Clinical Research Unit, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt Center for Human Nutrition, Nashville, Tennessee
  - Alchemi - Sugarland, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: Yes
Sharibg if protocol and ICF, pending FDA approval of this indication
Supporting Information: Study Protocol, ICF
Time Frame: Pending FDA Approval